CLINICAL TRIAL: NCT03675789
Title: Endotoxemia in Coronary Thrombus of Patients With Acute Coronary Syndrome
Brief Title: LPS and Platelet Activation in Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Francesco Violi, Director, Head of Internal Medicine, Clinical Professor, University of Roma La Sapienza
Other Study IDs: EMI-Sapienza
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
Keywords: Thrombi; LPS; Platelet Thrombus
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood, aspirated intra-coronary blood, aspirated coronary thrombi, aspirated plaque fragments from coronary culprit lesions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- STEMI: 50 STEMI patients treated with standard therapy undergoing to primary percutaneous coronary internention (PPCI). Thromboaspiration will be performed whenever possible (when the anatomy of the coronary artery - curve and size- allowed it) in all patients with a TIMI Flow 0 and in all patients with a visible thrombus if TIMI Flow was 1 or more.
- Stable angina: 50 stable angina (SA) patients on standard therapy, undergoing to intracoronary blood aspiration during elective diagnostic and/or interventional coronary procedure, matched for age, sex and comorbidities with the 50 STEMI patients.
- Controls: 50 outpatients without coronary heart disease, matched for age gender and comorbidities like diabetes and hypertension with the 50 STEMI patients. Peripheral blood samples will be collected during routine patient monitoring.

SUMMARY:
Platelets play a key role in the athero-thrombotic process. However, the in vivo mechanism accounting for thrombus growth at site of coronary atherosclerotic lesion has not been fully elucidated. While platelet adhesion and aggregation on the thrombogenic core of atherosclerotic plaque is an established mechanism for thrombus growth, the role of systemic factors, which may contribute to thrombus via amplification and propagation of platelet aggregation, is still to be clarified.

There is a growing body of evidence that lipopolysaccharides (LPS), are implicated in athero-thrombosis. Circulating levels of endotoxins have been associated with human atherosclerosis progression, particularly in smokers or in patients with infections. Furthermore, endotoxins seem to be implicated in the thrombotic process through several mechanisms including up-regulation of macrophage tissue factor expression and amplification of platelet response upon interaction with Toll-like receptor 4. The relationship between endotoxins and platelets may be relevant in the context of acute coronary syndromes as endotoxins could locally amplify platelet-derived thrombus growth but this issue is still unexplored.

Previous studies demonstrated that low-grade endotoxemia is detectable in human circulation, likely as consequence of enhanced gut permeability, and may be responsible for leucocyte-platelet aggregate and eventually thrombosis. The investigators hypothesize that low-grade endotoxemia may be observed in patients with coronary heart disease and may favor, at site of coronary unstable plaque, thrombus growth. To explore this issue, Escherichia Coli (EC)-LPS concentration and biomarkers of platelet activation will be measured in coronary thrombus and intra-coronary blood of patients with STEMI and stable angina (SA), respectively, and in peripheral circulation of both patients and controls. EC DNA will be searched in serum of all patients by polymerase chain reaction (PCR). Furthermore, to substantiate that LPS could be biologically active, immune-histochemical analysis of thrombi and in vitro studies will be performed to assess the interplay between LPS and platelet activation.

DETAILED DESCRIPTION:
In this case-control study, three groups of patients will be compared: consecutive STEMI patients undergoing to manual thrombo-aspiration during primary percutaneous coronary intervention, patients with chronic stable angina (SA) undergoing elective diagnostic and/or interventional coronary procedure and outpatients without coronary heart disease referring to the ambulatory of the Department of Internal Medicine, I Clinica Medica, Sapienza -University of Rome.

Patients will be recruited from three Centers: i) Department of the Heart and Great Vessels "Attilio Reale", Sapienza -University of Rome; ii) Department of Internal Medicine, I Clinica Medica, Sapienza -University of Rome; iii) Department of Interventional Cardiology, Santa Maria University Hospital, Terni.

The study complied with the Declaration of Helsinki and was approved by the local ethic committees of centers involved.

In patients presenting STEMI, coronary thrombi, when present, or plaque fragments will be aspirated from the culprit coronary artery before stent implantation and collected in EDTA tubes.

Thrombi will be homogenized in 5 mL of a homogenization buffer. Aliquots of thrombi homogenate will be centrifuged. In a subset of STEMI patients, part of the thrombotic material aspirated will be fixed in 4% buffered formaldehyde for histologic and immunohistochemical analyses.

In patients with SA, intracoronary blood will be aspirated from the stented coronary artery, before stenting, and immediately collected in EDTA tubes and centrifuged. Next, supernatant will be removed and stored at -80°C until use.

Peripheral blood samples will be obtained from a radial or femoral artery, before the start of procedure and after stent deployment in STEMI patients, or before balloon dilation and stenting in SA patients and then collected into tubes with or without 3.8% sodium citrate and EDTA tubes and centrifuged to obtain supernatant. Blood samples of controls group will be obtained from patients after supine rest for at least 10 min and taken into tubes with or without 3.8% sodium citrate and in EDTA tubes and centrifuged to obtain supernatant. Plasma and serum aliquots will be stored at -80°C in appropriate cuvettes until assayed.

Complete haemochrome, blood glucose, lipid profile, fibrinogen, creatinine, creatine kinase-MB and troponin T will be evaluated using standard methods.

sCD40L and sP-selectin levels will be measured with a commercial immunoassay in aliquots of plasma, thrombus homogenate and intracoronary blood.

Lipopolysaccharide (LPS) levels in serum and thrombus will be measured using a commercial ELISA kit.

A PCR reaction for specific amplification of a region of the 16S ribosomal RNA gene of Escherichia coli will be developed.

Serum zonulin levels will be measured using a commercial ELISA kit.

Immunoistochemistry (IHC) will be performed on sections obtained from formalin-fixed and paraffin embedded thrombus fragments aspirated from a subset of STEMI patients. After rehydration and antigen retrieval slides will be incubated with primary antibodies respectively to LPS, TLR4 and Cathepsin G, then washed in phosphate saline buffer and incubated with a secondary universal antibody. Immunoreactions will be detected with diaminobenzidine.

.

ELIGIBILITY:
Inclusion Criteria:

For STEMI patients:

* diagnosis of STEMI based on the current European Guidelines

For SA patients:

* diagnosis of SA defined according to the European Guidelines as lack of episodes of coronary instability for at least 6 months prior to admission

For control subjects:

* outpatients without diagnosis of coronary heart disease

Exclusion Criteria:

* estimated glomerular filtration rate less than 30 ml/min/m2
* acute or recent systemic infections (3 weeks)
* treatment with systemic corticosteroids
* treatment with oral anticoagulants
* malignancy
* lack of consent to participate

Additional exclusion criteria for STEMI patients were symptoms duration>12 h, rescue PCI, in-stent thrombosis and anatomical difficulty in reaching the lesion.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. STEMI patients referred to the catheterization laboratory for PPCI, who will undergo to manual coronary thrombo-aspiration, that fulfilled the inclusion/exclusion criteria, with a sufficient thrombotic material (≥1 mm3).
  2. patients with chronic stable angina (SA) undergoing elective diagnostic and/or interventional coronary procedure, undergoing to intracoronary blood aspiration
  3. outpatients without coronary heart disease matched for age, gender and comorbidities like diabetes and hypertension
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
LPS in blood of STEMI, SA patients and controls. | 1 year
  LPS will be measured in serum and expressed as concentration (pg/ml)

SECONDARY OUTCOMES:
LPS in thrombus and intra-coronary blood of STEMI and SA patients. | 1 year
  LPS will be measured in coronary thrombi of STEMI patients and in intra-coronary blood of SA patients and expressed as concentration (pg/ml)
sP-selectin in thrombus and intra-coronary blood of STEMI and SA patients. | 1 year
  sP-selectin (a marker of platelet activation) will be measured in coronary thrombi of STEMI patients and in intra-coronary blood of SA patients and expressed as concentration (ng/ml).
sCD40L in thrombus and intra-coronary blood of STEMI and SA patients. | 1 year
  sCD40L (a marker of platelet activation) will be measured in coronary thrombi of STEMI patients and in intra-coronary blood of SA patients and expressed as concentration (ng/ml).
Escherichia coli-DNA | 1 year
  Escherichia coli-DNA will be searched in serum patients and controls by polymerase chain reaction (PCR).The investigators will evaluate the rate of positivity in the serum of the study population.
Histologic and immunohistochemical analyses of thrombus fragments aspirated from a subset of STEMI patients. | 1 year
  Immunoistochemistry on sections obtained from formalin-fixed and paraffin embedded thrombus fragments.The investigators will analyze the composition of thrombus fragments and the presence of LPS , TLR4 and Cathepsin G.
HS-CRP in blood of STEMI, SA patients and controls | 1 year
  High sensitivity-C reactive protein will be measuer in serum and expressed as concentration (mg/L).
sP-selectin in blood of STEMI, SA patients and controls. | 1 year
  sP-selectin (a marker of platelet activation) will be measured in plasma and expressed as concentration (ng/ml)
Soluble CD40L (sCD40L) in blood of STEMI, SA patients and controls. | 1 year
  sCD40L (a marker of platelet activation) will be measured in plasma and expressed as concentration (ng/ml)
Zonulin in blood of STEMI, SA patients and controls | 1 year
  Zonulin (a marker of gut permeability) will be measued in serum and expressed as concentration (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — University of Roma La Sapienza
Locations (1):
- Internal and Medical Specialities Department - Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided